CLINICAL TRIAL: NCT02117882
Title: Minimally Invasive Lateral Approach for Sinus Augmentation: a Split-mouth Randomized Clinical Trial.
Status: Completed | Type: Observational
Sponsor: University of Firenze and Siena, Napoli, Italy (Other)
Responsible Party: Principal Investigator, nicola baldini, oral surgeon, University of Firenze and Siena, Napoli, Italy
Other Study IDs: misfe
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Bone Involvement in Diseases Classified Elsewhere
Keywords: lateral approach, bone augmentation , sinus floor elevation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- minimally invasive approach test: minimally invasive lateral approach
- control lateral traditional approach: standard surgical approach

SUMMARY:
It is assumed that the minimally invasive lateral approach and the traditional lateral sinus lift procedure will result in better outcomes in terms of height of augmented bone.

It is also assumed that the minimally invasive lateral approach will reduce surgical complications and patient's discomfort in comparison with a traditional lateral sinus lift procedure.

DETAILED DESCRIPTION:
16 patients edentulous in maxillary posterior area will be treated with a bilateral sinus lift procedure.

Once a patient will be enrolled in the study impressions will be taken. After the wax-up, a radiographic stent will be prepared. Special attention will be given to position radio-opaque references in the positions where the implants will be inserted according to a prosthodontic guided insertion. Pre-surgical CT scan will be executed after placing the stent in its proper position in patient's mouth. After that, if no surgical contra-indications will be detected at CT evaluation, patients will be enrolled for surgical interventions.

ELIGIBILITY:
Inclusion Criteria:

* - patient edentulous in the maxillary posterior area on both left and right side( not completely edentulous).
* - residual bone height in the maxillary premolar and molar region less than 4mm.

Exclusion Criteria:

* - history of systemic diseases that would contraindicate surgical treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 15 patients edentulous in maxillary posterior area have been treated with a bilateral sinus lift procedure.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
height of augmented bone | 6 months

SECONDARY OUTCOMES:
post surgical patient's discomfort | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: nicola nb baldini, oral surgeon, Principal Investigator — tuscan school of dental medicine of florence and siena
Locations (1):
- Siena University, Department of Periodontology, Policlinico Le Scotte Siena., Siena, Siena, Italy